CLINICAL TRIAL: NCT03769077
Title: Cycle to Fun - 'Exergames' for Inpatient Rehabilitation for Children/Youth With CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: Queen's University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB # 18-772
Record Dates: First submitted 2018-11-27; First posted 2018-12-07 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2018-11

CONDITIONS: Cerebral Palsy; Orthopedic Surgery
Keywords: Cerebral Palsy; Orthopedic Surgery; Exergames; Motor Function; Rehabilitation; GMFCS; Pain Reduction; Cycling
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergaming (Case) Group (Experimental): Participants assigned to the exergame condition will play the exergames for 30 minutes, 5 days a week for 3 weeks (15 exergame sessions). Outcomes will be acquired at baseline (before intervention), and at the end of every week during the 3 week intervention phase. Participants will also receive the current standard PT care at the Specialized Orthopedic and Developmental Rehab (SODR) inpatient unit at Holland Bloorview Kids Rehabilitation Hospital.
  The research participants will be asked to complete the following self-report questionnaires: Patient Reported Outcome Measurement Information System Pediatric Pain Interference Scale (PROMIS-PI), the KIDSCREEN-27, Faces Pain Scale-Revised (FPS-R) and the Self-Reported Experiences of Activity Settings (SEAS).
  Interventions: Device: Exergaming
- Comparison Group (No Intervention): Participants will receive the current standard PT care at the Specialized Orthopedic and Developmental Rehab (SODR) inpatient unit at Holland Bloorview Kids Rehabilitation Hospital and will complete questionnaires and assessments at the same time points during study participation.
  The research participants will be asked to complete the following self-report questionnaires: Patient Reported Outcome Measurement Information System Pediatric Pain Interference Scale (PROMIS-PI), the KIDSCREEN-27, Faces Pain Scale-Revised (FPS-R) and the Self-Reported Experiences of Activity Settings (SEAS).

INTERVENTIONS:
Device: Exergaming — This study involves the use of multiplayer exercise video games or 'exergames' that incorporate an avatar powered by pedaling a recumbent stationary bicycle. The Liberi suite of exergames contains six mini-games, including a combination of cooperative games, competitive games and individual games designed to be fast-paced, action-oriented, and enjoyable for youth with special needs.
  Arms: Exergaming (Case) Group

SUMMARY:
This study is designed to evaluate the feasibility and primary responses of a 3-week exergaming cycling program called Liberi Exergames for pediatric inpatients with cerebral palsy who are recovering from orthopedic surgery. This study involves the use of multiplayer exercise video games or 'exergames' that incorporate an avatar powered by pedalling a recumbent stationary bicycle. The Liberi suite of exergames contains six mini-games, including a combination of cooperative games, competitive games and individual games designed to be fast-paced, action-oriented, and enjoyable for youth with special needs. Standardized questionnaires and assessments investigating post-operative pain, gross motor function, quality of life, and study engagement are also administered. Five participants will engage in 'exergaming' sessions every weekday for 3 weeks, and five participants will only complete the assessments and questionnaires. All participants will receive the standard of care physiotherapy.

DETAILED DESCRIPTION:
As children with ambulatory CP become teenagers, they experience a decrease in their physical function and mobility. Many children/youth with CP develop contractures (i.e., shortening of their muscles) and bony deformities (e.g., hip subluxation) that require lower limb orthopedic surgery at some point between the ages of 7-16 years. Post-operatively this is followed by intensive rehabilitation to regain motor function. These youths often engage in sedentary activities and have low motivation to actively participate in physiotherapy thereby limiting their mobility, fitness, and overall well-being. Furthermore, pain is common during the post-surgical recovery period and is aggravated by muscle spasms.

Cycling is often incorporated into post-orthopedic rehabilitation programs in adults and has shown to reduce muscle spasms and improve range of motion post-hip replacement surgery. However, studies have yet to look at the role of cycling post-orthopedic surgery in youth with CP. Exercise video games or 'exergames' are a novel approach to engage youth with special needs in physical exercise and social interaction with their peers. To date the investigator's team of rehabilitation and computer scientists has developed an accessible and functional recumbent bicycling-based exergaming station, called the Liberi Exergames. These multiplayer exergames are designed to be fast-paced, action-oriented and enjoyable for youth with special needs and have been developed specifically for youth with CP.

The purpose of this case comparison study is to compare exergaming and standard physiotherapy to standard physiotherapy alone, in children with CP who are recovering from orthopedic surgery in an inpatient setting. This study is designed to evaluate the feasibility and primary responses to cycling with the Liberi Exergames. The primary outcomes are recruitment capability and acceptability as well as satisfaction of the intervention. Secondary outcomes are pain, health-related quality of life, and lower limb passive range of motion.

The first five participants will be recruited into the 'comparison' group and will participate in all study procedures except for the 'Exergaming' sessions. This will be followed by recruitment of 5 participants into the 'case' group, who will participate in the 'Exergaming' sessions as well as completing standardized assessments and questionnaires. All participants will receive physiotherapy as per standard of care.

Children/youth in the case group will play the Liberi Exergames for approximately 30 minutes per session in the afternoon, 5 days a week for three weeks. With the appropriate warm up/cool down, plus transfer on and off the unit, the total time for each training session will be approximately 45 minutes. The exergames will be supervised by a therapeutic recreation specialist and research staff, with transfers on and off the bike supervised by physiotherapy and/or nursing staff. The participants will not start the 3 week Exergame sessions until after they have started weight-bearing (i.e. for children who have received soft-tissue releases this is anticipated immediately post-operatively; for children who have had bony procedures this is anticipated at 4 weeks post-operatively).

Each exergaming station involves a specialized seat equipped with a seatbelt and lateral support that is connected to a MagneTrainer pedaling unit (3D Innovations, Greely, Colorado). The cycling unit is connected to a Toshiba DX730 computer. During the first session of the intervention, the bicycles will be fit to the participants by adjusting their length, the pedals, the position of the lateral supports, and their pedaling resistance.

The Liberi suite of exergames contains six mini-games, including a combination of cooperative games, competitive games and games that can be played individually. At the beginning of the 3 weeks training, research staff will make sure that the children/youth understand the games to be played. The participants will be situated in the same room when playing together. Participants will also wear a wireless heart rate (HR) monitor that can communicate with the gaming station using Bluetooth technology.

Participants will also be asked to complete questionnaires at the end of every week during the intervention phase. These assess post-operative pain (FPS-R, PROMS-PI), quality of life (KIDSCREEN-27), and activity engagement (SEAS) for all participants. A lower limb passive Range of Motion (PROM) will be conducted prior to the first exergaming session and after the final exergaming session. Participants will also be evaluated by the physiotherapist on their engagement in the standard of care physiotherapy sessions received by both groups (PRIME-O).

ELIGIBILITY:
Inclusion Criteria:

* Children/youth diagnosed with CP admitted to Holland Bloorview Kids Rehabilitation Hospital for inpatient rehabilitation following lower extremity orthopedic surgery
* Between 7 to 18 years of age
* Pre-operative Gross Motor Functional Classification Scale (GMFCS) level I - III
* Willingness and ability to operate a hand-held controller and pedal on the Liberi Exergames system
* Ability to self-report on the Faces Pain Scale-Revised (FPS-R)
* Documentation of informed consent by participant and/or representative and/or caregiver

Exclusion Criteria:

- Presence of unmanaged medical conditions (like exercise-induced asthma, heart condition, and uncontrolled seizures) that might prevent ability to train with the Liberi Exergames system

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
Percentage of eligible participants recruited [Feasibility] | 4 months
  Patients must meet all eligibility criteria in order to be included in the analysis of this outcome measure. A higher proportion of eligible patients recruited is considered to be a better outcome.
Percentage of participants who complete the Faces Pain Scale-Revised at baseline and at the end of the third week of the intervention phase [Feasibility] | End of week 3 of the intervention phase
  Good adherence with the assessments and outcome measures will be demonstrated if 100% of participants complete the FPS-R obtained at baseline and at the end of the third week of the intervention phase.
Percentage of participants who complete at least 12 of 15 Liberi Exergame Sessions [Feasibility] | End of week 3 of the intervention phase
  Adherence with the intervention protocol will aim for completion of >12 sessions out of 15 30-minute sessions administered over 3 weeks for each participant in the case group.

SECONDARY OUTCOMES:
Faces Pain Scale-Revised (FPS-R) | Baseline, end of weeks 1, 2, and 3 of the intervention phase
  The FPS-R is a faces scale used to obtain self-reported pain intensity scores. The FPS-R consists of six gender- and race-neutral faces portraying expressions from 'no pain' (scored "0") to 'very much pain' (scored "10") placed horizontally. The child is asked to point to the face that indicates how much pain she/he feels, and her/his reported pain is consequently scored using 2-point intervals (i.e., 0, 2, 4, 6, 8, and 10) for the six faces.
Patient Reported Outcome Measurement Information Systems Pediatric Pain Interference Scale (PROMIS-PI) | Baseline, end of weeks 1, 2, and 3 of the intervention phase
  The PROMIS-PI is an 8-item questionnaire that measures "pain interference" or the extend to which pain hinders physical, psychological, and socio-emotional functioning in daily activities. Each item has a five-option response scale ranging in value from 1 to 5, where '1=never' and '5=almost always'. All responses are summed to obtain a total raw score and score conversion tables are used to translate the total raw score into a T-score metric (mean= 50, standard deviation=10) for each participant. Higher scores indicate greater symptoms of pain or higher level of impairment.
KIDSCREEN-27 | Baseline, end of week 3 of the intervention phase
  The KIDSCREEN-27 is a globally used standardized health-related quality of life questionnaire measuring five Rasch scaled dimensions of wellbeing including: (1) Physical Well-being (5 items), (2) Psychological Well-being (7 items), (3) Autonomy and Parents (7 items), (4) Peers and Social Support (4 items), and (5) School Environment (4 items). Responses are indicated using a 5-point ordinal scale with responses ranging from 'never' to 'always', 'not at all' to 'extremely', or 'poor' to 'excellent'.
Change in Lower Limb Passive Range of Motion (PROM) | Baseline, end of week 3 of the intervention phase
  Passive range of motion of 16 joints will be recorded using standardized protocol and a universal goniometer. Hip flexion, extension, abduction, adduction, internal and external rotation of the hip, knee flexion and extension, and ankle dorsiflexion and plantar flexion will be measured bilaterally for each participant. Increased motion (as measured in degrees of rotation) is considered to be a better result.
Pediatric Rehabilitation Intervention Measure of Engagement-Observation (PRIME-O) | End of week 2 of the intervention phase
  The PRIME-O is a 10-item survey that asks the therapists to rate signs of engagement for the child/youths, themselves, and the child-PT interaction during therapy sessions. The PRIME-O is a tool developed for evaluating a child's engagement in pediatric rehabilitation interventions by capturing observations on three components of engagement: affective, cognitive and behavioral. The PRIME-O items are presented using a 5-point ordinal scale with responses ranging from '0 = Not at All' to '4 = To a Great Extent', with increased responses indicating increased interest and enthusiasm.
Self-Reported Experiences of Activity Settings (SEAS) | End of week 2 of the intervention phase
  The SEAS index is targeted toward children, including children with disabilities, and provides self-assessment of experience during an activity. Questions capture mood, enjoyment, sense of control, and sense of belonging within a group. Participants are asked to indicate agreement with a series of statements and responses are provided using a 7-point ordinal scale with responses ranging from 'Strongly Agree' to 'Strongly Disagree'.

CONTACTS AND LOCATIONS:
Overall Officials: Darcy Fehlings, MD, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada